CLINICAL TRIAL: NCT04402970
Title: Inhaled Dornase Alfa for Treatment of ARDS in Patients With SARS-CoV-2
Brief Title: Dornase Alfa for ARDS in Patients With Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV-2)
Acronym: DORNASESARS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Zach Holliday, Assistant Professor of Clinical Medicine, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022206
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV 2; ARDS
MeSH Terms: interventions — dornase alfa

STUDY DESIGN:
Intervention Model Description: Nebulized dornase alfa will be administered through the ventilator circuit at a dose of 2.5 mg, 12 hours apart, for 3 consecutive days. Patients will also receive lung protective ventilation (VC 6-8 ml/kg predicted body weight), plateau pressure < 30 centimeters of water pressure (cmH2O), targeted driving pressure < 15, neuromuscular blockade if indicated, and prone positioning based upon arterial blood content to fraction of inspired oxygen ratio (PaO2/FiO2) < 150 or upon treating physician decision; along with all other ICU care based upon best practice standards and evidence based medicine.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Inhaled/nebulized dornase alfa (Experimental): Patient to receive inhaled/nebulized dornase alfa (Pulmozyme) 2.5 mg twice daily in the ventilator circuit for 3 days, along with standard of care for ARDS.
  Interventions: Drug: Dornase Alfa Inhalation Solution
- Standard of care (No Intervention): Standard of care provided for ARDS.

INTERVENTIONS:
Drug: Dornase Alfa Inhalation Solution — Nebulized dornase alfa
  Other Names: Pulmozyme
  Arms: Inhaled/nebulized dornase alfa

SUMMARY:
This study is designed to evaluate a potential mechanism by which a hyperactive immune response may contribute to death from SARS-CoV-2; by an excessive neutrophil-mediated deposition of cell-free DNA in neutrophil extracellular traps (NET). Excessive amounts of NETs can increase rigidity of mucus, clog airways, and be agents for the development of acute respiratory distress (Narasaraju et al., Am J Pathol. 2011). Many aspects of this pathway have been observed in severe SARS-CoV-2 (Zhang et al., Respiratory research. 2020). Dornase alfa (DNAse I; Pulmozyme (Genentech) is a nebulized drug that works by degrading cell-free DNA and thus promoting airway clearance and recovery. The investigators hypothesize that by thinning mucus and degrading these NETs further lung damage may be prevented and a reduction in time to recovery may occur. The two aims of the study are to see if inhaled/nebulized dornase alfa will improve clinical outcome measures in SARS-CoV-2 related acute respiratory distress syndrome (ARDS) and to see if dornase alfa reduces the amount of bronchoalveolar lavage and blood markers of NET activity.

The study will recruit patients who are on mechanical ventilation for respiratory failure related to SARS-CoV-2 positive infection and have ARDS based upon Berlin criteria.

The investigators aim to recruit 10-20 patients for this study.

DETAILED DESCRIPTION:
Severe cases of SARS-CoV-2 infection have shown an inflammatory neutrophil and mucus-mediated airway exclusion pathway similar to previously described acute respiratory distress syndrome (ARDS) in other viral syndromes (Narasaraju et al., Am J Pathol. 2011). Lung neutrophilia in ARDS is related to significant neutrophil extracellular trap (NET) production and formation. Thus, NET production is likely contributing to the severe lung pathology in SARS-CoV-2 (Yu Zuo et al. Journal of Clinical Investigation Insight. 2020). Recent connections have been made between NET formation in SARS-CoV-2 patients and excessive thrombosis and the development of cytokine storm further warranting evaluation as a potential site for consideration of treatment (Barnes, Betsy et al. J exp Med. 2020). Dornase alfa (Pulmozyme) is a recombinant human deoxyribonuclease I, that acts as a mucolytic by cleaving extracellular chromosomal DNA from NETs and other cell-free DNA. Unknown are the effects of dornase alfa therapy on SARS-CoV-2 related ARDS and if therapy with dornase alfa truly reduces the amount of NETs in the severely damaged lungs.

This study is a non-randomized, single-center, open-label clinical trial to evaluate the potential benefit and cellular mechanism of nebulized dornase alfa administration in mechanically ventilated patients with SARS-CoV-2 related ARDS. Evaluation of dornase alfa effects at a cellular level will be measured by analysis of blood samples before and after the 3 days of therapy for cell-free DNA, quantification of citrullinated histone H3, quantification of Myeloperoxidase-DNA complexes and analysis of bronchoalveolar lavage samples for quantification of NETs and cell count and differential.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Hospitalized and mechanically ventilated for illness related to SARS-CoV-2
* Confirmed positive SARS-CoV-2 infection by Polymerase chain reaction (PCR)
* individual or surrogate ability to sign informed consent
* negative, urine-based pregnancy test in females

Exclusion Criteria:

* contraindication or intolerance to dornase alfa
* mechanical ventilation expected to be less than 48 hours
* life expectancy less than 24 hours based upon judgement of treating physician
* pregnant
* inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary M Holliday, MD, Principal Investigator — University of Missouri-Columbia; Adam Schrum, PhD, Study Director — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital and Clinics, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes BJ, Adrover JM, Baxter-Stoltzfus A, Borczuk A, Cools-Lartigue J, Crawford JM, Dassler-Plenker J, Guerci P, Huynh C, Knight JS, Loda M, Looney MR, McAllister F, Rayes R, Renaud S, Rousseau S, Salvatore S, Schwartz RE, Spicer JD, Yost CC, Weber A, Zuo Y, Egeblad M. Targeting potential drivers of COVID-19: Neutrophil extracellular traps. J Exp Med. 2020 Jun 1;217(6):e20200652. doi: 10.1084/jem.20200652. PMID 32302401
- [Background] Narasaraju T, Yang E, Samy RP, Ng HH, Poh WP, Liew AA, Phoon MC, van Rooijen N, Chow VT. Excessive neutrophils and neutrophil extracellular traps contribute to acute lung injury of influenza pneumonitis. Am J Pathol. 2011 Jul;179(1):199-210. doi: 10.1016/j.ajpath.2011.03.013. Epub 2011 May 7. PMID 21703402
- [Background] Zhang G, Zhang J, Wang B, Zhu X, Wang Q, Qiu S. Analysis of clinical characteristics and laboratory findings of 95 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a retrospective analysis. Respir Res. 2020 Mar 26;21(1):74. doi: 10.1186/s12931-020-01338-8. PMID 32216803
- [Background] Earhart AP, Holliday ZM, Hofmann HV, Schrum AG. Consideration of dornase alfa for the treatment of severe COVID-19 acute respiratory distress syndrome. New Microbes New Infect. 2020 Apr 30;35:100689. doi: 10.1016/j.nmni.2020.100689. eCollection 2020 May. PMID 32355564
- [Background] Zuo Y, Yalavarthi S, Shi H, Gockman K, Zuo M, Madison JA, Blair C, Weber A, Barnes BJ, Egeblad M, Woods RJ, Kanthi Y, Knight JS. Neutrophil extracellular traps in COVID-19. JCI Insight. 2020 Jun 4;5(11):e138999. doi: 10.1172/jci.insight.138999. PMID 32329756
- [Derived] Holliday ZM, Earhart AP, Alnijoumi MM, Krvavac A, Allen LH, Schrum AG. Non-Randomized Trial of Dornase Alfa for Acute Respiratory Distress Syndrome Secondary to Covid-19. Front Immunol. 2021 Oct 20;12:714833. doi: 10.3389/fimmu.2021.714833. eCollection 2021. PMID 34745093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-randomized 10 patients in inhaled dornase alfa arm and 20 patients in case-control (standard of care) arm
Groups:
- Standard of Care: Standard of care provided for Acute Respiratory Distress Syndrome (ARDS)
Period: Overall Study
Arm/Group | Inhaled/Nebulized Dornase Alfa | Standard of Care
Started | 10 | 20
Completed | 10 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled/Nebulized Dornase Alfa | Standard of Care | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Continuous [Mean (Full Range); unit: years] | 62 [47 to 79] | 58 [24 to 84] | 60 [24 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 6 | 13 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 8 | 16 | 24
  Black or African American | 0 | 1 | 1
  Hispanic or Latino | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 10 | 20 | 30
Diabetes mellitus [Count of Participants; unit: Participants] | 7 | 11 | 18
Hypertension [Count of Participants; unit: Participants] | 9 | 14 | 23
Coronary artery disease [Count of Participants; unit: Participants] | 5 | 7 | 12
Chronic lung disease (COPD, asthma, ILD) [Count of Participants; unit: Participants] | 3 | 7 | 10
Obesity [Count of Participants; unit: Participants] | 8 | 17 | 25
Remdesivir [Count of Participants; unit: Participants] — Received Remdesivir as therapy for Coronavirus disease 2019 (COVID-19)
  Participants | 9 | 20 | 29
Corticosteroids [Count of Participants; unit: Participants] — Received oral or intravenous corticosteroids as therapy for COVID-19
  Participants | 9 | 20 | 29
Antibiotics [Count of Participants; unit: Participants] — Received oral or intravenous antibiotics during hospital admission
  Participants | 10 | 19 | 29
Convalescent Plasma [Count of Participants; unit: Participants] — Received Convalescent Plasma therapy for COVID-19
  Participants | 9 | 11 | 20
Anticoagulation [Count of Participants; unit: Participants] — Received therapeutic dosing of anticoagulation during hospital admission
  Participants | 4 | 10 | 14
Paralytics [Count of Participants; unit: Participants] — Received paralytics during hospital admission
  Participants | 8 | 19 | 27
Prone positioning [Count of Participants; unit: Participants] — Treatment included prone positioning during hospital admission
  Participants | 8 | 16 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Arterial Blood Oxygen Content to Fraction of Inspired Oxygen Ratio (PaO2/FiO2)
Description: Daily evaluation of PaO2/FiO2 ratio at baseline prior to starting therapy and on days 1,2,3,4,5 and 14 if applicable
Time Frame: 14 days
Population: Number of patients still on mechanical ventilation and who underwent arterial blood gas monitoring to determine PaO2/FiO2 ratio
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Inhaled/Nebulized Dornase Alfa | Standard of Care
Number analyzed (Participants) | 10 | 20
mmHg
  Day 1 | 10.7 [-29.7 to 51.1] | 21.4 [-0.8 to 43.6]
  Day 2 | 61.1 [5.2 to 117] | 11.8 [-9.6 to 33.1]
  Day 3 | 23.5 [-21 to 68] | 12.5 [-9.7 to 34.7]
  Day 4 | 24.1 [-21.8 to 70.1] | 3.5 [-24.8 to 31.7]
  Day 5: number analyzed (Participants) | 8 | 20
  Day 5 | 37.6 [-35.9 to 111] | 5 [-28.8 to 38.8]
  Day 14: number analyzed (Participants) | 5 | 11
  Day 14 | 55 [-150.8 to 260.8] | -11.2 [-92.6 to 70.2]

2. Secondary Outcome: Change in Static Lung Compliance
Description: Daily evaluation of static lung compliance, measured by change in driving pressure over volume delivered, at baseline prior to starting therapy and on days 1,2,3,4,5 and 14 if applicable
Time Frame: 14 days
Population: Patients on mechanical ventilation with acute respiratory distress syndrome secondary to COVID-19
Measure: Mean (95% Confidence Interval); unit: mL/cmH20
Arm/Group | Inhaled/Nebulized Dornase Alfa | Standard of Care
Number analyzed (Participants) | 10 | 20
mL/cmH20
  Day 1: number analyzed (Participants) | 10 | 16
  Day 1 | 3.1 [-1.7 to 7.9] | -0.1 [-4.2 to 3.9]
  Day 2: number analyzed (Participants) | 10 | 15
  Day 2 | 4 [-1 to 9] | -0.4 [-3.1 to 2.3]
  Day 3: number analyzed (Participants) | 8 | 16
  Day 3 | 6.3 [-0.8 to 13.3] | -5.7 [-9.8 to -1.6]
  Day 4: number analyzed (Participants) | 8 | 15
  Day 4 | 4 [-3.2 to 11.3] | -5.6 [-9.4 to -1.8]
  Day 5: number analyzed (Participants) | 5 | 12
  Day 5 | 7.4 [-1.8 to 16.6] | -4.8 [-8.4 to -1.3]
  Day 14: number analyzed (Participants) | 4 | 6
  Day 14 | 0.8 [-16.3 to 17.8] | -10.2 [-17.9 to -2.4]

3. Secondary Outcome: Duration of Mechanical Ventilation
Description: Number of days on mechanical ventilation
Time Frame: From start of mechanical ventilation until extubation or date of death from any cause, whichever came first, assessed up to 6 months
Measure: Mean (Full Range); unit: Days
Arm/Group | Inhaled/Nebulized Dornase Alfa | Standard of Care
Number analyzed (Participants) | 10 | 20
Days | 15.2 [5 to 29] | 18.2 [8 to 38]

4. Secondary Outcome: Length of ICU Stay
Description: Number of days in the medical intensive care unit
Time Frame: From date of first admission to intensive care unit until discharge/transfer out of the ICU or date of death from any cause, whichever came first, assessed up to 6 months
Measure: Mean (Full Range); unit: Days
Arm/Group | Inhaled/Nebulized Dornase Alfa | Standard of Care
Number analyzed (Participants) | 10 | 20
Days | 16.5 [7 to 30] | 22.1 [11 to 47]

5. Secondary Outcome: Length of Hospitalization
Description: Number of days as an inpatient at the University of Missouri
Time Frame: From date of hospital admission until discharge from acute care hospital or date of death from any cause, whichever came first, assessed up to 6 months
Measure: Mean (Full Range); unit: Days
Arm/Group | Inhaled/Nebulized Dornase Alfa | Standard of Care
Number analyzed (Participants) | 10 | 20
Days | 22.5 [8 to 52] | 28.7 [15 to 60]

6. Secondary Outcome: Secondary Bacterial Infections
Description: Determination of secondary bacterial infections based upon positive culture results and clinical diagnosis by treating physician.
Time Frame: From date of randomization until first positive culture or clinical diagnosis of infection if occurs, assessed up to 3 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Inhaled/Nebulized Dornase Alfa | Standard of Care
Number analyzed (Participants) | 10 | 20
Percentage of participants | 30 [-5 to 65] | 25 [4 to 46]

7. Secondary Outcome: Mortality
Description: All cause mortality
Time Frame: 28 and 90 day evaluation
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Inhaled/Nebulized Dornase Alfa | Standard of Care
Number analyzed (Participants) | 10 | 20
Percentage of participants
  28 days | 40 [4 to 77] | 45 [21 to 69]
  90 days | 40 [4 to 77] | 55 [31 to 79]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected until end of hospitalization, death or up to 120 days whichever came first.
Description: Secondary pulmonary infections after the start of mechanical ventilation was the main adverse event data collected. Additional adverse events collected included development of blood stream infections or escalation of oxygenation support by need of extracorporeal membrane oxygenation therapy.
Arm/Group | Inhaled/Nebulized Dornase Alfa | Standard of Care
All-Cause Mortality (participants affected / at risk) | 4/10 | 11/20
Serious Adverse Events (participants affected / at risk) | 4/10 | 10/20
Other Adverse Events (participants affected / at risk) | 0/10 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled/Nebulized Dornase Alfa (N=10) | Standard of Care (N=20)
Bacteremia (Infections and infestations) | 1 (1) | 3 (3) — Development of blood stream infection after the start of mechanical ventilation
Ventilator associated pneumonia (Infections and infestations) | 3 (3) | 5 (5) — Development of ventilator associated pneumonia as determined by treating clinical physician
Venovenous extracorporeal membrane oxygenation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Need for escalation of respiratory support to venovenous extracorporeal membrane oxygenation support
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled/Nebulized Dornase Alfa (N=10) | Standard of Care (N=20)
Allergic reaction to drug (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Adverse reaction to inhaled dornase alfa including allergic reaction or acute need for escalation of oxygen therapy

LIMITATIONS AND CAVEATS:
Study was performed in non-randomized trial as there were initial concerns for low recruitment and difficulty with randomization. Study was also not powered for most secondary outcome analyses as it was designed in a pilot/feasibility status to determine drug effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT04402970/Prot_SAP_002.pdf
  • Informed Consent Form (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT04402970/ICF_004.pdf